CLINICAL TRIAL: NCT03632902
Title: Airway Management With Supraglottic Devices in Unruptured Intracranial Aneurysm Endovascular Therapy
Brief Title: Airway Management With Supraglottic Devices in Unruptured Intracranial Aneurysms
Status: Completed | Type: Observational
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Ricard Valero, head of neuroanesthesia section, Fundacion Clinic per a la Recerca Biomédica
Other Study IDs: HCB/2018/0691
Record Dates: First submitted 2018-06-26; First posted 2018-08-16 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Airway Management
Keywords: supraglottic devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: supraglottic device — airway management will be collected

SUMMARY:
Endovascular techniques for the treatment of intracranial aneurysms are growing.

DETAILED DESCRIPTION:
Retrospective analysis of the investigators experience in the last 8 years with the airway management in endovascular therapy for unruptured aneurysms. A total of 206 participants will be included from 2010 to 2018. Airway management (anticipated difficult airway, need for LM repositioning, orotracheal intubation because of failed laryngeal mask insertion, airway complication), intraoperative monitoring, aneurism size and location, intraoperative and perioperative complications will be registered.

Statistics will be compared between groups with t test or x test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent endovascular treatment for unruptured aneurysm

Exclusion Criteria:

* ruptured aneurysm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endovascular treatment for unruptured aneurysm in the past 8 years in our institution
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Security in the use of supraglottic devices in the unruptured intracranial aneurysms. | ten years
  security; the incidence of adverse events during the procedure and post-procedure will be recorded, also morbidity and mortality in patients managed with supraglottic devices during unruptured aneurysm embolization

CONTACTS AND LOCATIONS:
Overall Officials: PAOLA A HURTADO RESTREPO, md, Principal Investigator — anesthesiologist in Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No